CLINICAL TRIAL: NCT04027296
Title: Screening of COPD Patients at Risk of Complications in General Practice:
Brief Title: Development and Validation of the GLORI-COPD Score
Acronym: GLORI-COPD
Status: Active, not recruiting | Type: Observational
Sponsor: University of Paris 5 - Rene Descartes (Other)
Collaborators: Recherche Clinique Paris Descartes Necker Cochin Sainte Anne (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Alexandre MALMARTEL, Academic doctor of medicine, University of Paris 5 - Rene Descartes
Other Study IDs: 2018-A03259-46
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- suspected COPD: Patients aged ≥ 35yo and ≥10Pack.Year

SUMMARY:
The objective of this study is to evaluate the diagnostic accuracy of the GLORI-COPD score in ambulatory care, to enable the screening of COPD patients at risk of complications, requiring early management

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a chronic disease with a high prevalence in France, but which remains under-diagnosed due to the trivialization of symptoms and difficulty in accessing diagnostic investigations. It is associated with other co-morbidities, with an impact on the occurrence of complications and quality of life. Early management of the most severe patients would allow better control of these risks of complications. Our objective is to better identify patients with COPD at risk of complications in general practice, taking into account the totality of the patient, to improve their management.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 35 yo
* smoker or former smoker ≥ 10 Pack Years

Exclusion Criteria:

* Patients who have already been diagnosed with COPD by spirometry,
* have a contraindication to spirometry,
* have an estimated life expectancy of less than 5 years
* are under protective measures

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be any patient consulting a general practitioner over 35 years of age with smoking (active or weaned) in excess of 10 pack-years.
Sampling Method: Non-Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of the score | 12 months
  The diagnostic accuracy of the score will be evaluated to determine the risk of pulmonary complication in patients with COPD.
  Sensitivity, specificity, positive predictive value and negative predictive value

SECONDARY OUTCOMES:
COPD diagnosis | Baseline
  FEV1/FVC < 0.7
complications | 6 and 12 months
  -Composite criterion: Occurrence of a low respiratory infection (bronchitis, COPD exacerbation, lung infection or pneumonitis) in an outpatient or inpatient setting or following a death (1st event)
death | 12 months
Modified Medical Research Council Dyspnea scale score (mMRC) | baseline, 6 and 12 months
  evaluating dyspnea from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing
COPD Assessment test (CAT) | baseline, 6 and 12 months
  scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life
ADO index (Age, Dyspnea, Obstruction) | baseline, 6 and 12 months
  evaluates mortality risk in copd patients from 0 to 14 (higher scores are linked woh higher mortality risk)
GOLD stage | baseline
  COPD severity from A (less severe) to D (very severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Université Paris Cité, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malmartel A, Eap D, Ghasarossian C. [Spotting the GLObalRIsk of severe outcomes in undiagnosed COPD patients (GLORI-COPD)]. Rev Mal Respir. 2018 Mar;35(3):347-352. doi: 10.1016/j.rmr.2017.10.663. Epub 2018 Mar 27. French. PMID 29602483